CLINICAL TRIAL: NCT05326997
Title: Photobiomodulation With Yellow Light in the Treatment of Melasma: Clinical Trial, Randomized, Controlled, Double Blind.
Brief Title: Treatment of Melasma With Yellow Light Compared to Tranexamic Acid
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to implementation challenges, we categorized this study as a pilot and ended data collection, intending to adapt methods for future trials. Although the initial sample size was 54, data from 21 participants were analyzed.
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Christiane Pavani, Clinical Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRG
Record Dates: First submitted 2022-04-08; First posted 2022-04-14 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Melasma
Keywords: Low Level Laser Therapy (LLLT); Melasma; Photobiomodulation; Tranexamic Acid
MeSH Terms: conditions — Melanosis | interventions — Control Groups; Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: All participants will receive a skin preparation with enzymatic peeling, for homogeneity in the thickness of the stratum corneum among the participants and to reduce the unwanted reflection of photons. One week after the application of the peeling, the pre-treatment evaluation will be carried out and the participants will receive the intervention related to their treatment group, according to the allocation given by randomization. The area to be treated will be sanitized with Rennova® Beauté Micellar Water for makeup/sunscreen removal. Then, a cleaning foam based on 10% urea from Vivence laboratory will be used and also removed with gauze. After randomization, the study population will be divided into two groups (n=28 per group), wich are: (1) Group A - PBM with yellow LED application + placebo cosmetic treatment Home Care 2x per day, (2) Group B - PBM sham + treatment with 5% liposomal tranexamic acid Home Care cosmetic cream 2x per day.
Who Masked: Participant, Outcomes Assessor
Masking Description: Neither the participants involved in the study, nor the outcomes assessor will be aware of the groups formed, as well as the treatments received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation (PBM) with placebo cosmetic treatment. (Experimental): Participants will receive the intervention with PBM using amber light (DMC E-Light ABR), 20 J/cm² and will also receive a product for daily home topical use containing only the cosmetic base without active.
  Interventions: Device: Photobiomodulation group
- Photobiomodulation (PBM) sham with 5% liposomal tranexamic acid cosmetic product (Active Comparator): Participants will receive the simulated intervention with PBM using amber light (DMC E-Light ABR) and will also receive a product for topical home use containing 5% liposomal tranexamic acid.
  Interventions: Other: Group control (Tranexamic acid)

INTERVENTIONS:
Device: Photobiomodulation group — Participants will have their face sanitized with micellar water (a cosmetic product for cleaning and makeup remover), followed by cleaning with soap. Then, the eyes will be protected with gauze, proper glasses and a black towel on top, a headset with relaxation music will also be placed and then the face will receive the treatment with yellow light. After the session the face will receive sunscreen. A placebo cosmetic will be given to the participant to be applied twice a day and daily sunscreen.
  Arms: Photobiomodulation (PBM) with placebo cosmetic treatment.
Other: Group control (Tranexamic acid) — Participants will have their face sanitized with micellar water. Then, the eyes will be protected with gauze, proper glasses and a black towel on top, a headset with relaxation music will also be placed and then the face will receive the treatment with yellow light sham. The person responsible for applying the PBM will simulate the irradiations by positioning the device in the same places described for the PBM group, however, the equipment will be kept off. After the session the face will receive sunscreen. Will be delivered to patients, liposomal tranexamic acid with use 2 x a day home care and daily sunscreen.
  Arms: Photobiomodulation (PBM) sham with 5% liposomal tranexamic acid cosmetic product

SUMMARY:
Photobiomodulation (PBM) has been suggested as an alternative treatment for Melasma, showed by the in vitro data, inhibition of the tyrosinase enzyme and reduction in the pigment content by autophagy. This treatment compares with tranexamic acid, where it acts on similar pathways of melanogenesis. A total of 54 female participants, phototype scale Fitzpatrick ll - lV will be recruited which will be distributed among two groups: Light + placebo Home Care cosmetic product and Light sham + Home Care cosmetic product with tranexamic acid. The treatments will consist of 90 days, with application of photobiomodulation (PBM) once a week and application of the cosmetic product twice a day.

DETAILED DESCRIPTION:
This is a controled, randomized, double blind, two arms clinical trial. The main objective of this study is to evaluate the effect of photobiomodulation with amber light in the treatment of Melasma compared to the effect of tranexamic acid. The sample will be divided into 2 groups: Group 1 will receive PBM with amber Light Emitting Diode (LED) (DMC E-Light ABR), 20 J/cm² and placebo topical cosmetic for use in home care; Group 2 will receive PBM sham and topical cosmetic containing 5% liposomal tranexamic acid for use in home care. A total of 54 women with facial Melasma, aged 35 to 50 will be included. The treatments will consist of 12 sessions, once a week for 3 months. The severity of Melasma will be evaluated through the Melasma Area and Severity Index (MASI index), the pigmentation of the epidermis will be evaluated by corneomelametry, photographic records and the quality of life questionnaire (MELASQoL-PB) will also be made.

ELIGIBILITY:
Inclusion Criteria:

* Feminine gender
* Age between 35 to 50 years
* Phototypes l to lV of the Fitzpatrick scale
* Facial melasma
* Healthy participants without clinical skin comorbidities (psoriasis, vitiligo, rosacea and dermatoses)

Exclusion Criteria:

* Pre-existing systemic diseases, autoimmune diseases, digestive system disease
* Polycystic ovary
* Isotretinoin drug use (less than 6 months)
* Sequelae of an accident on the face that interferes with the facial treatment
* Undertakes any treatment for topical or oral Melasma at the time of the research or less than 3 months ago
* Uses retinoic acid, vitamin A derivatives, photosensitizing drugs
* Skin pathologies on the face
* Glaucoma, cataract, cancer patients, pregnant women, lactating women
* Uses oral or intrauterine contraceptives (IUD)
* Thyroid disorders
* Use of hormone replacement
* Bacterial, viral and fungal infections
* Tendency to form keloids

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
MASI (Melasma Area and Severity Index) | Before treatment (week 0).
  Determines the affected area and the severity of Melasma, through visual analysis of the affected site and attribution of scores
MASI (Melasma Area and Severity Index) | Half treatment (Week 6)
  Determines the affected area and the severity of Melasma, through visual analysis of the affected site and attribution of scores
MASI (Melasma Area and Severity Index) | After the treatments (week 12).
  Determines the affected area and the severity of Melasma, through visual analysis of the affected site and attribution of scores

SECONDARY OUTCOMES:
Corneomelametry | Before (week 0), at half (week 6) and after treatment (week 12).
  Quantifies the melanin present in the epidermis, specifically in the stratum corneum. A direct sample of the participant's skin will be collected with cyanoacrylate strippings (CSSS)
Photography | Before (week 0), at half (week 6) and after treatment (week 12).
  Registry of photographs at white and wood lamp
Final global diagnosis of the skin. | Before (week 0), at half (week 6) and after treatment (week 12).
  Clinical subjective measure with the aid of photographic records, in relation to the change by the severity of Melasma of pigmentation after treatment
The MELASQoL questionnaire, (Melasma Quality of Life Scale) | Before (week 0), at half (week 6) and after treatment (week 12).
  Evaluates the impact of Melasma on the quality of life of those affected by the disease and will be applied with the aim of evaluating facial self-image and their degree of satisfaction.
Adverse Effects | At half (week 6) and after treatment (week 12).
  Registry of any discomfort or unexpected effect of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thais Rodrigues Galache, MSc Fellow, Study Chair — University of Nove de Julho
Locations (2):
- Brazil (2):
  - Galache Clinic, São Caetano do Sul, São Paulo
  - Universidade Nove de Julho, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared. Researchers who provide a methodologically sound proposal will have access. Proposals should be directed to chrispavani@gmail.com To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Galache TR, Galache M, Barros RTB, Bezerra CDDS, Sena MM, Pavani C. Amber LED photobiomodulation versus tranexamic acid for the treatment of melasma: randomized controlled double-blind pilot trial. Lasers Med Sci. 2025 Jul 12;40(1):313. doi: 10.1007/s10103-025-04567-9. PMID 40650752
- [Derived] Galache TR, Galache M, Sena MM, Pavani C. Amber photobiomodulation versus tranexamic acid for the treatment of melasma: protocol for a double-blind, randomised controlled trial. BMJ Open. 2023 Jul 21;13(7):e073568. doi: 10.1136/bmjopen-2023-073568. PMID 37479524